CLINICAL TRIAL: NCT03876080
Title: Biomechanical Response to Dry Needling in Subjects With Delayed Onset Muscle Soreness: a Double Blind Randomized Control Trial
Brief Title: Dry Needling in Subjects With Delayed Onset Muscle Soreness
Acronym: TDNDOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley University (Other)
Responsible Party: Principal Investigator, Joseph Kelly, Assistant Professor, Bradley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CUHSR 71-18
Record Dates: First submitted 2019-02-05; First posted 2019-03-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Delayed Onset Muscle Soreness
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): Dry needling intervention to the gastrocnemius muscle trigger point
  Interventions: Other: Dry needling
- Sham needling (Sham Comparator): Sham dry needling intervention to the gastrocnemius muscle trigger point
  Interventions: Other: Sham needling

INTERVENTIONS:
Other: Dry needling — The use of a solid filiform needle to treat trigger points
  Arms: Dry needling
Other: Sham needling — Simulated needling
  Arms: Sham needling

SUMMARY:
Investigation of the biomechanical response in delayed onset muscle soreness using dry needling vs. sham

ELIGIBILITY:
Inclusion Criteria:

* The participants of the study will be any healthy male or female between
* age of 18 to 35
* able and willing to perform an exercise protocol using the gastrocnemius muscle
* willing to receive either sham or dry needling intervention

Exclusion Criteria:

* current muscular pain
* prior trigger point therapy in the past 6 months
* medications that affect muscle function
* injury in the past 6 months
* any health condition that prevents exercising
* recent surgery

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Change in Biomechanical stiffness (N/m) using MyotonPRO | baseline, immediately after intervention, 24 hours after intervention
  Measuring Biomechanical stiffness ( N/m) change at the following time frames

SECONDARY OUTCOMES:
Change in Pressure pain threshold using pressure algometry | baseline, immediately after intervention, 24 hours after intervention
  Measuring Pressure pain threshold change at the following time frames

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley University, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: No